CLINICAL TRIAL: NCT05578001
Title: Efficacy of Pilocarpine 1% in Pseudophakia Individuals With Presbyopia
Brief Title: Efficacy of Pilocarpine 1% in Presbyopia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Peyman, Dr. Alireza Peyman, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IR.MUI.MED.REC.1401.184
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Presbyopia; Pseudophakia
Keywords: Pilocarpine; Presbyopia; Pseudophakia
MeSH Terms: conditions — Presbyopia; Pseudophakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilocarpine (Experimental): 1 drop of Pilocarpine 1% instill in the eye
  Interventions: Drug: Pilocarpine Ophthalmic

INTERVENTIONS:
Drug: Pilocarpine Ophthalmic — 1 drop of Pilocarpine 1%
  Other Names: Glaupin 1%

SUMMARY:
In this before-after interventional study on patients with presbyopia after cataract surgery, uncorrected distance vision and corrected distance visual acuity are measured and recorded by Snellen chart. Corrected near visual acuity from a distance of 40 cm is measured by the standard near vision chart (Rosenbaum near vision card). Twenty minutes after the administration of pilocarpine 1%, the corrected near and far visual acuity is measured again. Also, the relationship between the difference in average near visual acuity after the administration of 1% pilocarpine in pseudophakic people is measured with iris color and pupil size.

DETAILED DESCRIPTION:
After selecting the study cases, the pupil size in both photopic and scotopic conditions and iris color(based on Simionescu's classification) will be recorded. Uncorrected distance visual acuity(UCDVA) will be measured by Snellen chart. Then the appropriate glasses will be placed according to the person's refraction and the corrected distance visual acuity(BCDVA) will be measured. Without changing the fitted glasses, corrected near visual acuity(BCNVA) is measured from a distance of 40 cm by the standard near vision chart (Rosenbaum near vision card). After this stage, one drop of pilocarpine 1% is prescribed in the patient's eye and 20 minutes later, the corrected near and far visual acuity is measured again. Thirty minutes and 8 hours after the administration of pilocarpine drop, the side effects of the drug, including headache, eye pain, eye redness, eye irritation, tearing, and blurred vision at night, are checked.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the study
* Previous uncomplicated cartaract surgery and PCIOL insertion
* BCDVA eqaul to or more than 8/10
* Less than 1.5 diopter cylindrical refractive error
* Spherical refractive error between -0.5_+1.5
* No history of previous eye disease
* Not using drugs that interact with pilocarpine

Exclusion Criteria:

* Occurrence of any drug-related complications
* Unable to follow up the patient after prescribing the drug

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Near Visual Acuity | 20 minutes
  Comparison of the BCNVA before and after instillation of Pilocarpine 1%

SECONDARY OUTCOMES:
Best Corrected Distance Visual Acuity | 20 minutes
  Comparison of the BCDVA before and after instillation of Pilocarpine 1%

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Peyman, M.D., Study Chair — Isfahan University of Medical Sciences, Isfahan, Iran
Locations (1):
- Isfahan Eye Research Center, Isfahan, Iran

REFERENCES:
- [Derived] Peyman A, Naderi-Lordejani M, Irajpour M, Ghanbarnia MJ, Koosha N, Pourazizi M. Pilocarpine 1% for Improved Near Vision in Pseudophakic Patients. J Ophthalmic Vis Res. 2025 May 19;20:10.18502/jovr.v20.15331. doi: 10.18502/jovr.v20.15331. eCollection 2025. PMID 40689127